CLINICAL TRIAL: NCT04623840
Title: Obesity-induced ED Response to Combined Effect of Tadalafil Drug in Addition to Interval and Continuous Training
Brief Title: Combined Effect of Continuous and Interval in Addition to Tadalafil Drug on Erectile Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, lecturer of Physical Therapy for Cardiovascular / Respiratory Disorder and Geriatrics, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/002918
Record Dates: First submitted 2020-11-04; First posted 2020-11-10 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercised group (Experimental): .(n=30) will be sedentary obese men with ED. All participants will receive five milligrams of tadalafil, one time per day, in addition to 3 sessions, per week, of combined continuous and interval aerobic exercise for eight weeks
  Interventions: Other: Tadalafil 5Mg Tab + continuous and interval exercise
- non-exercised group (Active Comparator): (n=30) will be sedentary obese men with ED. All participants will receive only five milligrams of tadalafil, one time per day, for eight weeks.
  Interventions: Drug: Tadalafil 5Mg Tab

INTERVENTIONS:
Other: Tadalafil 5Mg Tab + continuous and interval exercise — (n=30) will be sedentary obese men with ED. All participants will receive five milligrams of tadalafil, one time per day, in addition to 3 sessions, per week, of combined continuous and interval aerobic exercise for eight weeks
  Other Names: group 1
  Arms: Exercised group
Drug: Tadalafil 5Mg Tab — (n=30) will be sedentary obese men with ED. All participants will receive five milligrams of tadalafil, one time per day, for eight weeks
  Other Names: group 2
  Arms: non-exercised group

SUMMARY:
Erectile dysfunction (ED) is the persistent inability to attain and maintain a sufficient erection to permit satisfactory sexual performance. ED, a condition closely related to cardiovascular morbidity and mortality, is frequently associated with obesity. The importance of reducing cardiovascular risk factors remains fundamental to the overall vascular good health of the man, and that includes sexual vascular health. ED shares similar modifiable risks factors with coronary artery disease (CAD). Lifestyle modification that targets CAD risk factors may also lead to improvement in ED.

DETAILED DESCRIPTION:
Sixty obese men with ED complaints will be divided to two groups, exercised and non-exercised groups; n= 30 patients in every group. Both groups will receive five milligrams of tadalafil one time per day for 8 weeks but the exercised group only will receive - in addition to tadalafil - combined continuous and interval aerobic training, 3 session weekly for 8 weeks after detecting their target heart rate via the cardiopulmonary exercise test.

ELIGIBILITY:
Inclusion Criteria:

1. Sixty sedentary obese married men with BMI > 30 kg/m2.
2. The age of participants will range from 40-50 years old.
3. Blood pressure will be < 140/90 mm Hg.
4. The patients who will have ED at least from 6 months with IIEF-5 score < 22.

Exclusion Criteria:

1. Alcoholic, smoker, hypertensive, diabetic, and addicted patients.
2. Patients with pulmonary, renal, hepatic, and cardiac disorders.
3. Lower limb arthritis or orthopaedic disorders that will hinder the training program.
4. Prostatic inflammation, hyperplasia, and tumors.
5. Participation in a structured sport program in the previous 6 months.
6. previous pelvic and genital surgeries.

Ages: 40 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — self-representation of gender identity
Enrollment: 60 (Estimated)
Dates: Start 2020-10-12 (Actual); Primary Completion 2021-02-28 (Estimated); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
Five-Item Version of International Index of Erectile Function (IIEF-5) | It will be measured after eight weeks of training
  It is a questionnaire of five questions to diagnose ED in male patients

SECONDARY OUTCOMES:
Triglycerides | It will be measured after eight weeks of training
  It will be measured via a venous blood sample
High density lipoprotein | It will be measured after eight weeks of training
  It will be measured via a venous blood sample
Insulin | It will be measured after eight weeks of training
  It will be measured via a venous blood sample
Fasting blood glucose | It will be measured after eight weeks of training
  it will be measured via a blood glucose meter
The HOMA-IR (Homeostatic Model Assessment for Insulin Resistance | It will be measured after eight weeks of training
  HOMA-IR = [fasting insulin (μU/mL)
  × fasting glucose (mmol)]/22.5
body mass index | It will be measured after eight weeks of training
  It will be obtained by dividing the weight in Kilograms on the squared height in meter
systolic blood pressure | It will be measured after eight weeks of training
  it will be measured by a manual sphygmomanometer
diastolic blood pressure | It will be measured after eight weeks of training
  it will be measured by a manual sphygmomanometer
Waist circumference | It will be measured after eight weeks of training
  it will be measured by inelastic tape at the umbilicus level

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ismail, lecturer, Principal Investigator — Cairo University
Locations (1):
- Cairo Unoversity, Giza, Egypt